CLINICAL TRIAL: NCT06633471
Title: A Single-Center, Double- Masked, Randomized Study Evaluating the Safety and Efficacy of PS Therapy (PST) Tear Substitute Formulations in the Treatment of the Signs and Symptoms of Moderate Dry Eye Disease.
Brief Title: Clinical Study Aimed At Evaluating the Safety and Efficacy of Tear Substitute Formulations in the Treatment of Dry Eye Disease.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PS Therapy Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL001
Record Dates: First submitted 2024-10-01; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 30 subjects assigned to receive Rain (Experimental): Rain is one of the test formulations being evaluated for safety and efficacy in treating DED.
  Interventions: Drug: Two test formulations for the treatment of DED are being compared against the approved OTC formulation (Systane Ultra) and saline (placebo).
- 30 patients assigned to receive saline (Placebo Comparator): Saline is the placebo in this study.
  Interventions: Drug: Two test formulations for the treatment of DED are being compared against the approved OTC formulation (Systane Ultra) and saline (placebo).
- 30 subjects assigned to receive Mist (Experimental): Mist is one of the test formulations being evaluated for safety and efficacy in treating DED.
  Interventions: Drug: Two test formulations for the treatment of DED are being compared against the approved OTC formulation (Systane Ultra) and saline (placebo).
- 30 patients assigned to receive Systane Ultra (Active Comparator): Systane Ultra is the approved OTC formulation used to treat DED and the comparator for Rain and Mist.
  Interventions: Drug: Two test formulations for the treatment of DED are being compared against the approved OTC formulation (Systane Ultra) and saline (placebo).

INTERVENTIONS:
Drug: Two test formulations for the treatment of DED are being compared against the approved OTC formulation (Systane Ultra) and saline (placebo). — Rain and Mist are the test formulations. Systane Ultra is an approved OTC formulation. Saline is the placebo.

SUMMARY:
This clinical study is aimed at evaluating the safety and effectiveness of 2 test formulations (Rain and Mist), against an approved over-the-counter formulation (Systane Ultra) and a placebo (saline), in the treatment of moderate dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

Each subject must:

1. Be at least 18 years of age at the Screening Visit;
2. Of either gender and any race;
3. Be willing and able to follow all instructions and attend all study visits;
4. Have ALL of the following in the study eye1 at the Screening Visit:

   1. A corneal fluorescein staining score of ≥ 2 in at least one corneal region OR have a sum of ≥ 4 in all corneal regions
   2. A baseline Schirmer's Test (with topical anesthesia) Score of ≥ 2 millimeters (mm)/ and ≤ 10 mm/5 minutes
   3. A physician's diagnosis of Dry Eye Disease
5. Have normal lid/lash anatomy, blinking function and closure as determined by the Investigator;
6. Be literate and able to complete questionnaires independently;
7. Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug;
8. For females capable of becoming pregnant, agree to have urine pregnancy testing performed at screening (must be negative) and exit visits; must not be lactating; and must agree to use a medically acceptable form of birth control throughout the study. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months), or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).

Exclusion Criteria:

Each subject must not:

1. Have a known hypersensitivity to any of the procedural agents or study drug components, or have previously used the study drug;
2. Have clinically significant corneal epithelial defects at Visit 1, prior to performing Schirmer's Test;
3. Have had any intraocular surgery (such as cataract surgery) or extraocular surgery in either eye within three months, or refractive surgery (e.g., laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1;
4. Have had blepharoplasty in either eye;
5. Have had a corneal transplant in either eye;
6. Have used Restasis® or Xiidra® in the past 60 days;
7. Be using any ocular medications, other than the study treatment, within 7 days prior to Visit 1 and throughout the study treatment period. This includes both therapeutic and lubricant eye drops that could potentially interfere with the study outcomes, by either exacerbating or alleviating the symptoms of dry eye disease.
8. Have used contact lenses within 7 days prior to Visit 1 or anticipate the use of contact lenses during the study treatment period;
9. Have any form of punctal or intracanalicular occlusion;
10. Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with DED are allowed;
11. Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study, or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.);
12. Have active or uncontrolled, severe:

    * Systemic allergy
    * Chronic seasonal allergies at risk of being active during the study
13. Have any condition or history that, in the opinion of the Investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject;
14. Be currently enrolled in an investigational drug or device study, or have used an investigational drug or device within 30 days prior to Visit 1 and during the treatment period;
15. Be a female who is currently pregnant, planning a pregnancy or lactating.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Schirmer's Test | 4 weeks
  Mean change in Schirmer's Test Score (STS) from pre-instillation of IP to 5 minutes post-instillation of IP at Visits 1 and 2
Tear Film Break Up Time (TFBUT) | 4 weeks
  Mean change in Tear Film Break Up Time (TFBUT) from baseline to post- instillation of IP at each of Visits 1 and 2
Corneal Fluorescein Staining | 4 weeks
  Mean change from Baseline in Corneal Fluorescein Staining at Visits 1 and 2
Conjunctival Staining | 4 weeks
  Mean change from Baseline in Conjunctival Staining at Visits 1 and 2
Ocular Redness | 4 weeks
  Ocular redness, as evaluated by the Investigator, at Baseline at Visits 1 and 2 (0-4 unit scale, allowing half unit increments) assessed pre-dose at each visit

SECONDARY OUTCOMES:
Secondary Efficacy Parameters | 4 weeks
  Measurement of inflammatory markers using ELISA: Changes in the levels of specific inflammatory markers will be evaluated using Enzyme-Linked Immunosorbent Assay (ELISA) at specified timepoints (Visit 1 and 2) to assess the anti-inflammatory efficacy of the PST Tear formulations.
Adverse Events | 4 weeks
  Adverse Event (AE) Query
Slit Lamp Findings | 4 weeks
  Slit Lamp Biomicroscopy
IOP | 4 weeks
  Intraocular Pressure (IOP)
Fundoscopy | 4 weeks
  Dilated Fundoscopy

OTHER OUTCOMES:
Tolerability Measures | 4 weeks
  Drop comfort assessment (0-10 unit scale) assessed by subject immediately upon instillation, at 1 minute, 3 minutes, and 5 minutes post-instillation at Visit 1 and Visit 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Warrens Eye Care Centre, Bridgetown, Barbados